CLINICAL TRIAL: NCT03520270
Title: Potentially Inappropriate Treatments in Turkish ICUs: Point Prevalence Study
Brief Title: Prevalence of Potentially Inappropriate Treatments
Acronym: INAPPT-ICU
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, ELIF ERDOGAN, Principal Investigator, Istanbul University
Other Study IDs: EERDOGAN
Record Dates: First submitted 2018-04-13; First posted 2018-05-09 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Critical Illness; Terminal Illness; Potentially Inappropriate Medication List
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multicenter point prevalence study in Turkish intensive care units.

DETAILED DESCRIPTION:
Intensive care units (ICU) are life-saving units for critical patients with using advanced technology. In some cases, it becomes a unit where treatment is not possible, the fatal patients are admitted and the death process is extended. Most patients with end-stage cancer, advanced-stage chronic obstructive pulmonary disease (COPD) and advanced-stage Alzheimer's disease prefer to die at home, although many often refer to emergency services at the end of their life and are then transferred to the ICU. Intensive care treatments are often very invasive and painful interventions. The patient who lives in intensive care unit is faced with many psychological distresses such as communication, isolation and fear besides physical ache. For this reason, it is necessary to make decisions (end-of-life decisions) such as forbearing intensive care treatments applied to the patients in the death process or cutting out the ones started. In the world, the goal for the end of life patients is, improving the last phase of their lives with the application of these decisions and symptom therapy, living in a peace without pain and respiratory distress. However, there is an uncertanity in these issues in our country and intensive care physicians are hesitant to make decisions about the end of life with concern about legal problems. Although it is known that these patients will not benefit most from the treatment of ICU, they are getting treatments for saving their lives in ICUs. The fact that intensive care beds are not available due to the patients who are not get beneficial treatment, brings the result of difficult finding of the beds which will benefit from the intensive care, and in fact it is a waste of intensive care resources which is very expensive. The size of the problem is not known as there is no data on the frequency of patients in our country who are in intensive care and require end-of-life care.

In this multicenter point prevalence study our aims are;

* to find out the incidence of patients in intensive care units in Turkey in the last period of life,
* to compare the resource use of end-of-life and non-end-of-life patients.

ELIGIBILITY:
Inclusion Criteria:

All patients who are over 18 years old, more than 48 hours in the intensive care unit, or expected to be hospitalized

Exclusion Criteria:

Patients under 18 years of age, less than 48 hours in the intensive care unit stay, or who are monitorized for post-operative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All intensive care patients fulfilling eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of terminal patients in the ICU | 1 day
  Investigation of the number of terminal patients treated in the intensive care units at the last days of life

SECONDARY OUTCOMES:
Resource use | 1 day
  Comparison of treatment implementations such as antibiotics, use of mechanical ventilation, renal replacement therapy, nutrition and blood transfusions and their estimated costs, used for terminal and non-terminal patients

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa Medical School, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nelson JE, Bassett R, Boss RD, Brasel KJ, Campbell ML, Cortez TB, Curtis JR, Lustbader DR, Mulkerin C, Puntillo KA, Ray DE, Weissman DE; Improve Palliative Care in the Intensive Care Unit Project. Models for structuring a clinical initiative to enhance palliative care in the intensive care unit: a report from the IPAL-ICU Project (Improving Palliative Care in the ICU). Crit Care Med. 2010 Sep;38(9):1765-72. doi: 10.1097/CCM.0b013e3181e8ad23. PMID 20562699
- [Result] Shreves A, Marcolini E. End of life/palliative care/ethics. Emerg Med Clin North Am. 2014 Nov;32(4):955-74. doi: 10.1016/j.emc.2014.07.010. Epub 2014 Sep 16. PMID 25441045